CLINICAL TRIAL: NCT05727904
Title: A Phase 3, Multicenter, Randomized, Open-label, Parallel Group, Treatment Study to Assess the Efficacy and Safety of the Lifileucel (LN-144, Autologous Tumor Infiltrating Lymphocytes [TIL]) Regimen in Combination With Pembrolizumab Compared With Pembrolizumab Monotherapy in Participants With Untreated, Unresectable or Metastatic Melanoma
Brief Title: Study to Investigate Lifileucel Regimen Plus Pembrolizumab Compared With Pembrolizumab Alone in Participants With Untreated Advanced Melanoma.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Iovance Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IOV-MEL-301; TILVANCE-301 (Other: Iovance Biotherapeutics, Inc.); TILVANCE (Other: Iovance Biotherapeutics, Inc.)
Expanded Access: NCT05398640 (Available)
Record Dates: First submitted 2023-02-06; First posted 2023-02-14 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Melanoma; Unresectable Melanoma; Melanoma
Keywords: Tumor Infiltrating Lymphocytes; TIL; Metastatic Melanoma; Unresectable Melanoma; Cell Therapy; Cellular Immuno-therapy; IL-2; Non-myeloablative lymphodepletion (NMALD); Check point inhibitor; Melanoma; Lifileucel; Stage III Melanoma; Stage IV Melanoma; Skin cancer; Skin cancer types; Malignant melanoma; Autologous Adoptive Cell Therapy; Autologous Adoptive Cell Transfer; LN-144; Pembrolizumab; Pembro; Adjuvant/Neo-adjuvant; BRAF/MEK; ICI; BRAF v600; Immune checkpoint inhibitor; Tumor infiltrating T-cells; TILVANCE; TILVANCE-301
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — lifileucel; pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Lifileucel plus Pembrolizumab
  Interventions: Biological: Lifileucel plus Pembrolizumab
- Arm B (Active Comparator): Pembrolizumab alone with Optional Crossover Period
  Interventions: Biological: Pembrolizumab with Optional Crossover Period

INTERVENTIONS:
Biological: Lifileucel plus Pembrolizumab — A tumor sample is resected from each patient for Lifileucel manufacturing. Patients then receive Pembrolizumab followed by the lifileucel regimen which consists of non-myeloablative lymphodepletion, lifileucel infusion followed by IL-2. Patients will then continue to receive Pembrolizumab every 6 weeks until disease progression.
  Other Names: LN-144; Pembrolizumab
  Arms: Arm A
Biological: Pembrolizumab with Optional Crossover Period — Patient will receive Pembrolizumab monotherapy every 6 weeks until disease progression. Upon verified confirmed disease progression by the blinded independent review central committee, patients may proceed to lifileucel monotherapy during an optional crossover period if they meet eligibility criteria.
  Optional crossover: A tumor sample is resected from each patient for Lifileucel manufacturing. Patients then receive the lifileucel regimen which consists of non-myeloablative lymphodepletion, lifileucel infusion followed by IL-2.
  Arms: Arm B

SUMMARY:
This is a Phase 3, multicenter, open-label, randomized, parallel group, treatment study to assess the efficacy and safety of lifileucel in combination with pembrolizumab compared with pembrolizumab alone in participants with untreated, unresectable or metastatic melanoma. Participants randomized to the pembrolizumab monotherapy arm who subsequently have a blinded independent central review- verified confirmed progressive disease (PD) will be offered lifileucel monotherapy in an optional crossover period.

DETAILED DESCRIPTION:
The study will enroll participants with unresectable or metastatic melanoma (Stage IIIC, IIID, or IV per the American Joint Committee on Cancer [AJCC] staging system) who have had no prior therapy for metastatic disease. Previous adjuvant/neoadjuvant therapy with a single line of protooncogene B-Raf (BRAF) inhibitor with or without a mitogen-activated protein kinase (MEK) inhibitor, PD-1 inhibitor, or cytotoxic T-lymphocyte-associated antigen-4 [CTLA-4] inhibitor is allowed, provided such treatment was completed ≥6 months before progression to metastatic disease.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has a histologically or pathologically confirmed diagnosis of Stage IIIC, IIID, or IV unresectable or metastatic melanoma.
2. In the investigator's assessment, the participant has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 and an estimated life expectancy of > 6 months.
3. Participant is assessed as having at least one resectable lesion (or aggregate lesions) for lifileucel generation.
4. Participant must have at least one measurable disease as defined by RECIST 1.1 following tumor resection.
5. Participants must have adequate organ function.
6. Participants of childbearing potential or those with partners of childbearing potential must be willing to practice an approved method of highly effective birth control.
7. Participants who are > 70 years of age may be allowed to enroll after the investigator discusses with the medical monitor.

Exclusion Criteria:

1. Participant has melanoma of uveal/ocular origin.
2. Participant has symptomatic untreated brain metastases.
3. Participant received more than 1 prior line of therapy.
4. Participant received prior therapy for metastatic disease
5. Participants with a BRAF V600 mutation-positive tumor received prior adjuvant/neoadjuvant ICI therapy only
6. Participant has an active medical illness(es) that, in the opinion of the investigator, would pose increased risks for study participation, such as systemic infections; seizure disorders; coagulation disorders; or other active major medical illnesses of the cardiovascular, respiratory, or immune systems.
7. Participant has any form of primary or acquired immunodeficiency (eg, SCID or AIDS).
8. Participant had another primary malignancy within the previous 3 years (except for those that do not require treatment or were curatively treated >1 year ago, and in the judgment of the investigator do not pose a significant risk of recurrence.)
9. Participant has a history of allogeneic cell or organ transplant.

Other protocol defined inclusion/exclusion criteria could apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 670 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate and Progression Free Survival | 5 years total duration
  To compare the efficacy of lifileucel plus pembrolizumab with the efficacy of pembrolizumab alone measured by objective response rate (ORR) and progression-free survival (PFS) assessed by the blinded independent review committee (BIRC) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1

SECONDARY OUTCOMES:
Overall Survival | 7 years total duration
  To compare the efficacy of lifileucel plus pembrolizumab with the efficacy of pembrolizumab alone measured by overall survival (OS)
Complete Response Rate, Duration of Response and Event Free Survival | 5 years total duration
  To compare the efficacy of lifileucel plus pembrolizumab with the efficacy of pembrolizumab alone measured by complete response (CR) rate and duration of response (DOR) and event- free survival (EFS) assessed by the BIRC per RECIST v1.1
Objective Response Rate, Progression Free Survival, Complete Response Rate, Duration of Responses, Event Free Survival and PFS2 | 5 years total duration
  To compare the efficacy of lifileucel plus pembrolizumab with the efficacy of pembrolizumab alone measured by ORR, PFS, CR rate, DOR, and EFS assessed by the investigator per RECIST v1.1 and PFS2 assessed by the investigator
Adverse Events | 5 years total duration
  To characterize the safety and tolerability profile of lifileucel plus pembrolizumab and pembrolizumab alone in participants with unresectable or metastatic melanoma

CONTACTS AND LOCATIONS:
Overall Officials: Iovance Biotherapeutics Study Team, Study Director — Iovance Biotherapeutics
Locations (72):
- United States (22):
  - University of Alabama at Birmingham: The Kirklin Clinic, Birmingham, Alabama
  - City of Hope, Duarte, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - California Pacific Medical Center, San Francisco, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Orlando Health Cancer Institute, Orlando, Florida
  - University of Illinois Hospital & Health Sciences System, Chicago, Illinois
  - University of Kansas, Kansas City, Kansas
  - University of Louisville - James Graham Brown Cancer Center, Louisville, Kentucky
  - National Cancer Institute, Bethesda, Maryland
  - Barbara Ann Karmanos Cancer Hospital dba Karmanos Cancer Center, Detroit, Michigan
  - Henry Ford Health, Detroit, Michigan
  - Dartmouth-Hitchcock Medical Center (DHMC) - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - MD Anderson Cancer Center at Cooper, Camden, New Jersey
  - Oncology Hematology Care, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - St. Luke's Cancer Center - Anderson, Easton, Pennsylvania
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Baptist Cancer Center, Bartlett, Tennessee
  - SCRI Oncology Partners, Nashville, Tennessee
  - Virginia Commonwealth University, Richmond, Virginia
  - Swedish Cancer Institute, Edmonds, Washington
- Australia (5):
  - Greenslopes Private Hospital, Greenslopes, Queensland
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Flinders Medical Centre, Bedford Park
  - Westmead Hospital, Westmead
- Universitair Ziekenhuis Brussel - Oncologisch Centrum, Jette, Belgium
- Canada (2):
  - Centre hospitalier de l'Université de Montréal, Montreal, Quebec
  - Princess Margaret Cancer Centre, Toronto
- France (3):
  - Institut Paoli Calmettes, Marseille
  - Centre Hospitalier Universitaire de Nantes (CHU de Nantes) - Hotel-Dieu, Nantes
  - Hopital Saint Louis, Paris
- Germany (4):
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Schleswig-Holstein - Campus Lübeck, Lübeck
  - Klinikum Rechts der Isar der Technischen Universität München, Munich
- Israel (3):
  - Hadassah Medical Center, Jerusalem
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (6):
  - Istituto Romagnolo per lo Studio dei Tumori, Meldola, Forlì-Cesena
  - Centro di Riferimento Oncologico IRCCS, Aviano, Friuli Venezia Giulia
  - Azienda Ospedaliero Universitaria Pisana, Pisa, Tuscany
  - Istituto Europeo Di Oncologia, Milan
  - Istituto Nazionale Per Lo Studio E La Cura Dei Tumori Fondazione Giovanni Pascale, Napoli
  - Azienda Ospedaliera Universitaria Senese, Siena
- Nederlands Kanker Instituut, Amsterdam, Netherlands
- South Korea (3):
  - Bundang Medical Center - CHA University, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (14):
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Regional Universitario de Malaga - Hospital General, Málaga, Málaga
  - Instituto Oncologico Rosell, Barcelona
  - Hospital Universitari Vall dHebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - ICO l'Hospitalet - Hospital Duran i Reynals, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitario Madrid Sanchinarro - CIOCC, Madrid
  - Hospital Universitario Quirónsalud Madrid, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Clínica Universitaria de Navarra, Pamplona
  - Hospital Universitario Virgen Macarena, Seville
  - Consorcio Hospital General Universitario de Valencia, Valencia
- Sahlgrenska Universitetssjukhuset, Gothenburg, Västra Götaland County, Sweden
- Centre Hospitalier Universitaire Vaudois Lausanne, Lausanne, Switzerland
- United Kingdom (6):
  - Queen Elizabeth Hospital Birmingham, Birmingham, England
  - Freeman Hospital, Newcastle upon Tyne, England
  - Royal Marsden Hospital, Chelsea, London
  - Beaston West of Scotland Canter Centre, Glasgow
  - Guy's Hospital, London
  - Sarah Cannon Research Institute UK, London